CLINICAL TRIAL: NCT04076904
Title: Cesarean Niche Examination by us to Assess Its Integrity and Dehescence
Brief Title: Cesarean Niche Examination by Transvaginal us
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher , lecturer ,Obstetrics and Gynecology , National Research Centre, Aljazeera Hospital
Other Study IDs: cesarean niche
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transvaginal us with 2D and 3D SHG — transvaginal us is made to all women with SHG

SUMMARY:
The developed uterine scar developing due to cesarean section is usually clinically evaluated and visualized by transvaginal sonography (TVS) and saline infusion sonography (SIS) or Gel installation sonography (GIS)

DETAILED DESCRIPTION:
In 2015, WHO displayed and reveled a systematic review of the research studies in the scientific literature to evaluate and asses the linkage and connection between cesarean section rates and maternal

ELIGIBILITY:
Inclusion Criteria:

- women with secondary infertility

Exclusion Criteria:

* obstructed labor, pregnant women having chronic diseases;

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females with a previous section and has secondary infertility
Study Population: In 2015, WHO displayed and reveled a systematic review of the research studies in the scientific literature to evaluate and asses the linkage and connection between cesarean section rates and maternal,
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
The number of women who will have dehesent scar | within a week
  transvaginal us showing lower segment with assessing scar

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (2):
- Egypt (2):
  - Algazeerah and Kasralainy hospital, Giza
  - Algazeerah, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alalfy M, Osman OM, Salama S, Lasheen Y, Soliman M, Fikry M, Ramadan M, Alaa D, Elshemy S, Abdella R. Evaluation of the Cesarean Scar Niche In Women With Secondary Infertility Undergoing ICSI Using 2D Sonohysterography Versus 3D Sonohysterography and Setting a Standard Criteria; Alalfy Simple Rules for Scar Assessment by Ultrasound To Prevent Health Problems for Women. Int J Womens Health. 2020 Nov 3;12:965-974. doi: 10.2147/IJWH.S267691. eCollection 2020. PMID 33177887